CLINICAL TRIAL: NCT00713219
Title: Phase II Study of Docetaxel + Cetuximab + Concurrent Re-Irradiation (Intensity -Modulated Radiation Therapy, IMRT) for Patients With Locoregionally Recurrent Head and Neck Cancer
Brief Title: Docetaxel + Cetuximab + Concurrent Re-Irradiation (Intensity - Modulated Radiation Therapy, IMRT) for Patients With Locoregionally Recurrent Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Oncology/Hematology West (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-050
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Results first posted 2015-04-23 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Head and Neck Cancer
Keywords: IMRT; cetuximab; docetaxel
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Cetuximab; Docetaxel

ARMS (1):
- 1 (Experimental): CHEMORADIATION
  Interventions: Radiation: IMRT, cetuximab, docetaxel

INTERVENTIONS:
Radiation: IMRT, cetuximab, docetaxel — IMRT will be administered in once daily fractions (2 Gy/day, Monday through Friday) over approximately 7 weeks to a goal of approximately 70 Gy. The chemotherapy regimen will begin with a loading dose of intravenous cetuximab (400 mg/m2) one week prior to the initiation of radiation therapy, followed by weekly administration of intravenous docetaxel (15 mg/m2) and intravenous cetuximab (250 mg/m2) for approximately 7 weeks concurrently with radiation. Patients will be evaluated weekly prior to their chemotherapy. All patients will be evaluated on an intention-to-treat basis.

SUMMARY:
This is a study for patients who have head and neck cancer that has recurred in the body area where they previously received radiation, and for whom surgery is not planned. A widely accepted treatment option in this situation is chemotherapy alone. Another approach that has been used in clinical trials is to treat patients with a repeat course of radiation. In these studies, some patients received chemotherapy at the same time as the radiation.

In this clinical study, we wish to treat with radiation plus two drugs during the course of reirradiation, Taxotere® (docetaxel) and Erbitux® (cetuximab). Docetaxel and cetuximab both are chemotherapy drugs which are administered by vein. Both drugs help radiation kill cancer cells.

The radiation will be administered using a strategy called intensity-modulated radiation therapy (IMRT), which focuses the radiation beam on the tumor.

Docetaxel and cetuximab are both approved for the treatment of patients with head and neck cancer.

However, the combination of radiation + docetaxel + cetuximab for patients with recurrent head and neck cancer is considered to be a topic for clinical research. The purpose of this study is to determine the good and bad effects of treatment with radiation + docetaxel + cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) confirmed diagnosis of recurrent or second primary head and neck squamous cell carcinoma (HNSCC) in patients with past history of definitive radiation therapy for head and neck cancer. Patients in whom the initial diagnosis was neck metastasis with suspected occult primary in the head and neck will be eligible.

Patients with histologic variants such as spindle cell carcinoma, poorly-differentiated keratin positive carcinoma, and lymphoepithelioma will be eligible.

* Patients may be eligible if they have unresected recurrent disease in the prior radiation field. Patients also may be eligible if they have undergone surgical resection of recurrent disease in the prior radiation field with any of the following poor risk pathologic features:

  * Malignant involvement of 2 or more regional lymph nodes
  * Extracapsular extension of nodal disease
  * Microscopically involved mucosal margins of resection (at 5 mM or less)
  * Perineural involvement
  * Resected soft tissue disease
  * Oral cavity or oropharyngeal primaries with nodal disease at levels IV or V
* Patients must have had prior radiation for head and neck cancer with ≥ 50 % of the recurrent tumor within areas that have been radiated to at least 45 Gy, but not exceeding 72 Gy.
* Greater than 6 month interval from prior external beam radiation treatment. (Patients who have received intra-operative radiation therapy [IORT] within 6 months of registration may be eligible, if there has been no subsequent disease recurrence in the IORT field and criteria for eligibility are otherwise met).
* KPS > or = to 70%
* Age > or = to 18years
* Adequate bone marrow function: ANC > or = to 1,500/μl, platelets > or = to 100,000/μl, Hgb > or = to 8 g/dL.
* Adequate hepatic function.
* Women of childbearing potential must have a negative pregnancy test.
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least three months thereafter.
* Patient must sign an informed consent document.

Exclusion Criteria:

* Anticipated lifetime spinal cord dose exceeding 54 Gy, brain stem exceeding 65 Gy, optic chiasm exceeding 55 Gy, and optic nerves exceeding 60 Gy.
* Three or more palliative cytotoxic chemotherapy regimens in the recurrent or metastatic disease setting.
* Pregnancy or lactation.
* Distant metastatic disease.
* Other active malignancy, other than indolent malignancies which the investigator determines are unlikely to interfere with treatment or efficacy analysis. For example, patients with nonmelanoma skin cancer, in situ carcinoma of the cervix, or prostate cancer within the no current biochemical (PSA) or radiologic evidence of disease may enroll.
* Serious concomitant medical disorders (for example, active infection, uncontrolled seizure disorder, unstable angina) that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study.
* History of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate-80.
* History of severe infusion reaction to a monoclonal antibody.
* Patients with multifocal peripheral sensory alterations or paresthesias (including tingling) interfering with function, per patient report (example: activities of daily living).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Fury, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Oncology/Hematology West, Omaha, Nebraska
  - Memorial Sloan-Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan-Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel + Cetuximab + Concurrent Re-Irradiation: Docetaxel + Cetuximab + Concurrent Re-Irradiation (Intensity - Modulated Radiation Therapy, IMRT) for Patients with Locoregionally Recurrent Head and Neck Cancer
Period: Overall Study
Arm/Group | Docetaxel + Cetuximab + Concurrent Re-Irradiation
Started | 14
Completed | 12
Not Completed | 2
Not completed — Death | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel + Cetuximab + Concurrent Re-Irradiation
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Progression-Free Survival (PFS).
Description: Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measureable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: conclusion of the study
Measure: Mean (Full Range); unit: Days
Arm/Group | Docetaxel + Cetuximab + Concurrent Re-Irradiation
Number analyzed (Participants) | 12
Days | 370 [91 to 1186]

ADVERSE EVENTS:
Arm/Group | Docetaxel + Cetuximab + Concurrent Re-Irradiation
Serious Adverse Events (participants affected / at risk) | 7/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel + Cetuximab + Concurrent Re-Irradiation (N=14)
Dehydration (General disorders) | 2 (2)
Syncope (fainting) (General disorders) | 2 (2)
Ocular/Visual - Other (specify) (Ear and labyrinth disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Allergic reaction (including drug fever) (General disorders) | 1 (1)
Infection unknown ANC-Pneumonia(lung) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage, Oral cavity (General disorders) | 1 (1)
Infection, other (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel + Cetuximab + Concurrent Re-Irradiation (N=14)
Constipation (Gastrointestinal disorders) | 2 (2)
Dehydration (General disorders) | 1 (1)
Dysphagia (Difficulty swallowing) (General disorders) | 1 (1)
Edema: limb (General disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3 (6)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 3 (5)
Glucose, low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2 (3)
Lymphopenia (Blood and lymphatic system disorders) | 10 (13)
Mucositis (Clinical exam)- Oral cavity (General disorders) | 4 (4)
Mucositis (symptoms)- Oral cavity (General disorders) | 2 (2)
Ocular/Visual (Eye disorders) | 1 (1)
Pain (General disorders) | 3 (3)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (2)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash: dermatitis associated with Chemoradiation (Skin and subcutaneous tissue disorders) | 3 (3)
Rash: dermatitis associated with Radiation (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes